CLINICAL TRIAL: NCT00171704
Title: A Study to Evaluate the Effect of Letrozole and Tamoxifen on Bone and Lipids in Postmenopausal Women With Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Collaborators: Danish Breast Cancer Cooperative Group (Other); University of Sheffield (Other)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CFEM345D2407
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Results first posted 2012-06-04 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2012-05

CONDITIONS: Hormone Sensitive Resected Primary Breast Cancer in Postmenopausal Women
Keywords: Breast Cancer; Letrozole; Bone Mineral Density; Bone Markers; Serum lipid; Postmenopausal
MeSH Terms: conditions — Breast Neoplasms | interventions — Letrozole; Tamoxifen

ARMS (2):
- Letrozole (Experimental): 2.5 mg once daily (q.d.)orally for 5 years
  Interventions: Drug: Letrozole
- Tam-Let (Experimental): 20 mg Tamoxifen once daily (q.d.) orally for 2 years followed by Letrozole 2.5 mg q.d. orally for 3 years.
  Interventions: Drug: Letrozole; Drug: Tamoxifen

INTERVENTIONS:
Drug: Letrozole — 2.5 mg tablets and supplied in bottles with 6-monthly supplies.
Drug: Tamoxifen — 20 mg tablets in bottles as 6-monthly supplies (supplied to Novartis as Tamofen from Schering Oy, Subsidiary of Schering AG, Pansiontie 47, FIN-2010 Turku, Finland)
  Arms: Tam-Let

SUMMARY:
Estrogen is known to be a regulator of bone and lipid metabolism. Letrozole is a potent inhibitor of estrogen synthesis.

This study evaluated the effects of letrozole and tamoxifen on bone and lipid metabolism in postmenopausal women with resected, receptor positive early breast cancer.

ELIGIBILITY:
Inclusion Criteria

* Female
* Post-menopausal hormone status defined as:
* Patients with menostasis (amenorrhea) > 12 months or history of oophorectomy.
* Patients ≥ 55 years with history of hysterectomy or having continued/renewed menstruation on cyclic hormone treatment.
* Patients of 50-54 years: Menopausal status was determined on the basis of follicle-stimulating hormone (FSH)/luteinizing hormone (LH) values.
* Histologically confirmed resected breast cancer and eligible for adjuvant endocrine therapy. As a minimum, patients had to have receptor-positive tumors, which were defined either as estrogen receptor (ER) and/or progesterone receptor (PgR) ≥ 10 fmol/mg cytosol protein; or ≥ 10% of the tumor cells positive by immunocytochemical evaluation.
* Adequate bone marrow function (white blood cell count [WBC] > 3.0 x 109 /L, platelets ≥ 100.0 x 109 /L, and hemoglobin > 10 g/dL).
* Documented evidence of adequate renal function (creatinine < 180 µmol/L) and hepatic function (bilirubin < 30 µmol/L, alanine aminotransferase (ALT) < 1.5 x upper normal limit of the laboratory).
* Life expectancy of at least 24 months at the time of enrollment.
* Written voluntary informed consent prior to initiation of any study procedure.
* Willingness to undergo all scheduled tests and examinations for evaluation of bone density and bone metabolism, and lipid profiles in addition to the standard assessments for monitoring their breast cancer status.

Exclusion Criteria

* Patients with distant metastases as defined by the criteria of the Danish Breast Cancer Co-operative Group (DBCCOG).
* Pre-existing bone disease (e.g. osteomalacia, osteogenesis imperfecta, Paget's disease).
* Patients receiving bisphosphonates for more than 3 months before randomization.
* Chronic treatment with drugs known to interfere with bone metabolism, e.g.
* Anti-convulsants within the past year.
* Corticosteroids at doses greater than the equivalent of 5 mg/day prednisone for more than two weeks in the past 6 months (prior to randomization).
* Any previous treatment with sodium fluoride at daily doses ≥ 5 mg/day for a period exceeding 1 month.
* Anabolic steroids in the past 12 months.
* Long term use of coumarin derivatives and heparin at the time of randomization.
* Metabolic diseases known to interfere with bone metabolism (e.g., Hyperparathyroidism, hypoparathyroidism, uncontrolled thyroid disease, Cushing's disease, vitamin D deficiency, malabsorption syndrome, etc.).
* Treatment with lipid-lowering agents within the 3 months prior to randomization (this exclusion criterion did not apply to patients randomized in the United Kingdom).
* Patients receiving other anti-cancer treatment.
* Previous neoadjuvant / adjuvant chemotherapy and /or previous adjuvant endocrine therapy (e.g., anti-estrogens, AIs).
* History of previous or concomitant malignancy within the past 5 years other than adequately treated basal or squamous cell carcinoma of the skin or in situ carcinoma of the cervix. Patients who had a previous other malignancy must have been disease free for five years. Patients with endometrial cancer and/or invasive breast cancer at any time in their medical history were excluded. Patients with invasive bilateral breast cancer were excluded. Patients with vaginal discharge/ vaginal bleeding with evidence of malignancy were excluded.
* Any other non-malignant systemic diseases (cardiovascular, renal, hepatic, lung embolism, etc.) which would prevent prolonged follow-up.

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 263 (Actual)
Dates: Start 2005-04; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Chair — Novartis
Locations (13):
- Denmark (12):
  - Novartis Investigative Site, Aalborg
  - Novartis Investigative Site, Aarhus
  - Novartis Investigative Site, Copenhagen
  - Novartis Investigative Site, Esbjerg
  - Novartis Investigative Site, Herlev
  - Novartis Investigative Site, Herning
  - Novartis Investigative Site, Hillerød
  - Novartis Investigative Site, Kløvervænget
  - Novartis Investigative Site, Roskilde
  - Novartis Investigative Site, Sønderborg
  - Novartis Investigative Site, Vejle
  - Novartis Investigative Site, Viborg
- Novartis Investigative Site, Sheffield, United Kingdom

RESULTS

PARTICIPANT FLOW:
Groups:
- Tam-Let: Tamoxifen 20 mg once daily (q.d.) orally for 2 years followed by Letrozole 2.5 mg q.d. orally for 3 years.
Period: Overall Study
Arm/Group | Letrozole | Tam-Let
Started | 133 | 130
Completed | 89 | 81
Not Completed | 44 | 49
Not completed — Adverse Event | 24 | 33
Not completed — Disease Progression | 14 | 9
Not completed — New therapy for 2nd non-breast prim canc | 1 | 0
Not completed — Administrative Problems | 2 | 1
Not completed — Death | 2 | 2
Not completed — Withdrawal by Subject | 1 | 3
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Letrozole | Tam-Let | Total
Number analyzed (Participants) | 133 | 130 | 263
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.4 (6.1) | 61.8 (6.2) | 61.6 (6.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 133 | 130 | 263
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline of Bone Mineral Density of the Lumbar Spine (L2-l4)
Description: Lumbar spine (L2-L4) BMD measurements by dual energy X-ray absorptiometry (DXA) were performed after surgery and within 2 weeks prior to randomization and repeated every 6 months for the first 2 years and annually thereafter until 5 years after enrollment. The primary scanning site was the lumbar spine (L2 to L4) and the secondary scanning site was the total hip. All DXA scans were evaluated by a central reader.
Time Frame: Baseline, 24 months
Population: The safety population consisted of only patients who took randomized therapy for at least one day. The number of patients in each treatment arm who had completed 2 years of the study and had centrally assessed measurements of lumbar spine or total hip BMD.
Measure: Median (Full Range); unit: Percent Change
Arm/Group | Letrozole | Tam-Let
Number analyzed (Participants) | 63 | 68
Percent Change | -4.63 [-14.21 to 4.32] | 0.37 [-6.98 to 15.21]

2. Secondary Outcome: Percent Change From Baseline of Bone Mineral Density of the Lumbar Spine
Description: Lumbar spine (L2-L4)BMD measurements by dual energy X-ray absorptiometry (DXA) were performed after surgery and within 2 weeks prior to randomization and repeated every 6 months for the first 2 years and annually thereafter until 5 years after enrollment. The primary scanning site was the lumbar spine (L2 to L4) and the secondary scanning site was the total hip. All DXA scans were evaluated by a central reader.
Time Frame: Baseline, 60 months
Population: The safety population consisted of only patients who took randomized therapy for at least one day. The analysis at 5 years included all patients enrolled and who had centrally assessed measurements of lumbar spine and/or total hip BMD.
Measure: Median (Full Range); unit: Percent change
Arm/Group | Letrozole | Tam-Let
Number analyzed (Participants) | 56 | 53
Percent change | -5.66 [-15.06 to 5.11] | -3.3 [-13.48 to 4.92]

3. Secondary Outcome: Percent Change From Baseline of Bone Mineral Density (BMD) of Total Hip
Description: Total hip BMD measurements by dual energy X-ray absorptiometry (DXA) were performed after surgery and within 2 weeks prior to randomization and repeated every 6 months for the first 2 years and annually thereafter until 5 years after enrollment. All DXA scans were evaluated by a central reader.
Time Frame: Baseline, 60 months
Population: The safety population consisted of only patients who took randomized therapy for at least one day. The analysis of BMD at 5 years included all patients enrolled with centrally assessed measurements of total hip BMD.
Measure: Median (Full Range); unit: Percent Change
Arm/Group | Letrozole | Tam-Let
Number analyzed (Participants) | 62 | 65
Percent Change | -5.77 [-22.53 to 12.53] | -3.98 [-13.6 to 5.57]

4. Secondary Outcome: Median Percent Change From Baseline of Serum Markers of Bone Turnover
Description: Bone turnover markers (fasting serum procollagen-I extension peptide [P1NP], C-telopeptide [CTX], skeletal bone-specific alkaline phosphatase [BSAP, N-telopeptide [NTX]) were measured at baseline/screening and at each visit thereafter. A central laboratory was used to analyze the samples. The analysis of bone markers was based on analysis of variance of the regression slopes calculated for each individual patient and each bone marker over time. In the following summary, only the median treatment group percent change from baseline (and range) at 5 years is presented for each bone marker.
Time Frame: Baseline, 60 months
Population: The safety population consisted of only patients who took randomized therapy for at least one day. During different time points, participants with observations at that time point were included in the analysis. The analysis of bone markers over time consisted of patients with measurements of specific markers at each time point.
Measure: Median (Full Range); unit: Percent Change
Arm/Group | Letrozole | Tam-Let
Number analyzed (Participants) | 133 | 130
Percent Change
  Procollagen-I (PINP) (n=86, 78) | -14.15 [-78.5 to 177.8] | -0.5 [-84.8 to 200]
  Bone Specific alkaline Phosphatase (n=87,78) | 16.2 [-53.6 to 192.6] | 19.15 [-58.00 to 237.8]
  C-telopeptide (CTX) (n=88, 78) | -12.05 [-80.9 to 130.6] | 4.55 [-81.2 to 236.8]
  N-telopeptide (NTX) (n=-88, 77) | -53.05 [-86.3 to 20.2] | -50.7 [-100 to 39]

5. Secondary Outcome: Percentage Change From Baseline in Serum Lipids at 5 Years
Description: Serum lipid profile (fasting serum cholesterol [total, HDL and calculated LDL], triglycerides, and lipoprotein [a]) were measured at baseline/screening and at each visit thereafter. A central laboratory was used to analyze the samples. The analysis of serum lipids was on the treatment group median percent change from baseline (and range) at 5 years.
Time Frame: Baseline, 60 months
Population: The safety population consisted of only patients who took randomized therapy for at least one day. During different time points, participants with observations at that time point were included in the analysis.
Measure: Median (Full Range); unit: Percent Change
Arm/Group | Letrozole | Tam-Let
Number analyzed (Participants) | 133 | 130
Percent Change
  Total Cholesterol (n=91, 82) | -7.3 (17.64) [-45.2 to 34.7] | -2.45 (16.63) [-55.7 to 24.5]
  LDL Cholesterol (n=91, 82) | -12.7 (24.947) [-63.9 to 58.3] | -11.05 (23.958) [-65 to 48.4]
  HDL Cholesterol (n=91, 82) | 8.7 (16.388) [-40 to 60] | 8.9 (-38.5) [-38.5 to 68.8]

6. Secondary Outcome: Number of Participants With Clinically Relevant Changes From Baseline in Cholesterol
Description: Serum lipid profile (fasting serum cholesterol [total, HDL and calculated LDL], triglycerides, and lipoprotein [a]) were measured at baseline/screening and at each visit thereafter. A central laboratory was used to analyze the samples. Numbers are not additive, as patients could be included in multiple rows.
Time Frame: Baseline, 60 months
Population: The safety population consisted of only patients who took randomized therapy for at least one day. The number of patients with pre-defined clinically relevant changes in serum lipids over the course of 5 years in each treatment arm is presented.
Measure: Number; unit: Participants
Arm/Group | Letrozole | Tam-Let
Number analyzed (Participants) | 133 | 130
Participants
  Patients with one or more change | 30 | 21
  ≥8 mmol/L total (T) cholesterol | 7 | 5
  ≥7 mmol/L T.choles. & ≥1 risk for cardiac disease | 18 | 12
  ≥6 mmol/L T. choles. & ≥2 risk for cardiac disease | 11 | 9

7. Secondary Outcome: Time to Disease Recurrence or Death
Description: Disease-free survival was defined as the interval between randomization and earliest confirmed event of loco-regional recurrence, distant metastases, invasive contralateral breast cancer, or death from any cause.
Time Frame: 60 months
Population: Analysis of disease-free survival was based on the ITT principle, with all enrolled (and randomized) patients included. The Kaplan-Meier product-limit approach was used.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Letrozole | Tam-Let
Number analyzed (Participants) | 133 | 130
Days | NA [NA to NA] — Median time to disease recurrence or death was not achieved, nor was it possible to estimate 25% or 75th percentile for disease free survival. | NA [NA to NA] — Median time to disease recurrence or death was not achieved, nor was it possible to estimate 25% or 75th percentile for disease free survival.

8. Secondary Outcome: Time to Overall Survival Events
Description: Overall survival was measured from date of randomization to date of death.
Time Frame: 60 Months
Population: All randomized patients constituted the ITT Population, unless withdrawal of consent occurred after randomization but before the start of study treatment assigned.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Letrozole | Tam-Let
Number analyzed (Participants) | 133 | 130
days | NA [NA to NA] — Median time to death was not achieved; nor was it possible to estimate 25th or 75th percentile for overall survival. | NA [NA to NA] — Median time to death was not achieved; nor was it possible to estimate 25th or 75th percentile for overall survival.

ADVERSE EVENTS:
Groups:
- Letrozole: 2.5 mg once daily q.d. orally for 5 years
Arm/Group | Letrozole | Tam-Let
Serious Adverse Events (participants affected / at risk) | 50/133 | 41/130
Other Adverse Events (participants affected / at risk) | 113/133 | 110/130
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Letrozole (N=133) | Tam-Let (N=130)
Acute myocardial infarction (Cardiac disorders) | 0 | 2
Angina pectoris (Cardiac disorders) | 1 | 1
Angina unstable (Cardiac disorders) | 0 | 1
Arrhythmia (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 2 | 2
Atrial flutter (Cardiac disorders) | 0 | 1
Bundle branch block left (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1
Pericarditis (Cardiac disorders) | 0 | 1
Sinus bradycardia (Cardiac disorders) | 0 | 1
Goitre (Endocrine disorders) | 1 | 0
Retinal detachment (Eye disorders) | 2 | 0
Abdominal hernia (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Diverticulum (Gastrointestinal disorders) | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Medical device complication (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 1
Breast infection (Infections and infestations) | 0 | 2
Bronchitis (Infections and infestations) | 0 | 1
Cystitis (Infections and infestations) | 0 | 1
Diverticulitis (Infections and infestations) | 3 | 0
Encephalitis herpes (Infections and infestations) | 1 | 0
Erysipelas (Infections and infestations) | 1 | 2
Herpes zoster (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 4 | 1
Skin infection (Infections and infestations) | 2 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 2 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 2 | 1
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 0
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 1 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 5 | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Benign breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Benign salivary gland neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Breast cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Gastrooesophageal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hypopharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Thyroid adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebral infarction (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 2
Dizziness (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 0
Calculus ureteric (Renal and urinary disorders) | 1 | 0
Colpocele (Reproductive system and breast disorders) | 2 | 0
Cystocele (Reproductive system and breast disorders) | 0 | 1
Ovarian cyst (Reproductive system and breast disorders) | 1 | 0
Rectocele (Reproductive system and breast disorders) | 0 | 1
Uterine polyp (Reproductive system and breast disorders) | 1 | 0
Uterine prolapse (Reproductive system and breast disorders) | 1 | 1
Uterovaginal prolapse (Reproductive system and breast disorders) | 0 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Scar (Skin and subcutaneous tissue disorders) | 0 | 1
Skin irritation (Skin and subcutaneous tissue disorders) | 1 | 0
Social problem (Social circumstances) | 1 | 0
Social stay hospitalisation (Social circumstances) | 0 | 1
Breast reconstruction (Surgical and medical procedures) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 2
Hypotension (Vascular disorders) | 0 | 1
Orthostatic hypotension (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Letrozole (N=133) | Tam-Let (N=130)
Constipation (Gastrointestinal disorders) | 11 | 6
Nausea (Gastrointestinal disorders) | 14 | 12
Fatigue (General disorders) | 7 | 15
Oedema peripheral (General disorders) | 17 | 15
Radiation skin injury (Injury, poisoning and procedural complications) | 6 | 10
Weight decreased (Investigations) | 6 | 7
Weight increased (Investigations) | 5 | 7
Hypercholesterolaemia (Metabolism and nutrition disorders) | 23 | 21
Arthralgia (Musculoskeletal and connective tissue disorders) | 44 | 43
Back pain (Musculoskeletal and connective tissue disorders) | 14 | 25
Bone pain (Musculoskeletal and connective tissue disorders) | 16 | 10
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 11 | 8
Myalgia (Musculoskeletal and connective tissue disorders) | 5 | 12
Osteopenia (Musculoskeletal and connective tissue disorders) | 15 | 12
Osteoporosis (Musculoskeletal and connective tissue disorders) | 21 | 8
Pain in extremity (Musculoskeletal and connective tissue disorders) | 13 | 5
Headache (Nervous system disorders) | 3 | 7
Depression (Psychiatric disorders) | 6 | 12
Insomnia (Psychiatric disorders) | 5 | 8
Vaginal discharge (Reproductive system and breast disorders) | 15 | 12
Vulvovaginal dryness (Reproductive system and breast disorders) | 10 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 8
Alopecia (Skin and subcutaneous tissue disorders) | 7 | 6
Hot flush (Vascular disorders) | 13 | 18
Hypertension (Vascular disorders) | 25 | 17
Lymphoedema (Vascular disorders) | 7 | 2

LIMITATIONS AND CAVEATS:
The study was designed to investigate the effects of letrozole compared with tamoxifen for 2 years on BMD spine (L2-L4). The study was too small to investigate the comparative efficacy of treatments on disease-free survival or on overall survival.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal Investigators are NOT employed by the organization sponsoring the study. Other disclosure agreement that restricts the right of the PI to discuss or publish trial results after the trial is completed. The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in clinical trial.